CLINICAL TRIAL: NCT02140177
Title: Ask Suicide-Screening Questions to Everyone in Medical Settings (asQ'em): Development of a Suicide Risk Screening Instrument for Adult Medical Inpatients
Brief Title: Ask Suicide-Screening Questions to Everyone in Medical Settings (asQ em): Development of a Suicide Risk Screening Instrument for Adult Medical Inpatients
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140109; 14-M-0109
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Questionnaires and Surveys
Keywords: Screening; Adults; Medical Inpatients; Suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Adult Medical Inpatients: Adult medical inpatients; We will enroll adult patients, ages 18 years and older, admitted to identified inpatient medical units during designated data collections days.

SUMMARY:
Background:

- Suicide is the 10th leading cause of death for U.S. adults. Medically ill people are at an increased risk of suicide. Most people who have killed themselves went to a healthcare provider within 3 months of their death. More and more, hospitals are being asked to assess people for signs of suicide risk so that they can get the help they need. If nurses and doctors can find out who is at risk they can make sure these people get help in the hospital.

The asQ em (Ask Suicide-Screening Questions to Everyone in Medical Settings) is a brief questionnaire. It was created to detect suicidal thoughts and behaviors in hospitalized people. Researchers would like to further develop this tool and figure out which are the best questions to ask patients.

Objective:

- To determine the best questions for healthcare providers to ask people with medical illnesses to see if they are having suicidal thoughts or planning to hurt themselves.

Eligibility:

- NIH Clinical Center patients over age 18.

Design:

* Participants will be asked questions about how they have been feeling in the past few weeks. They will be asked questions about depression, anxiety, and suicidal thoughts and behaviors. They also will be asked some background questions.
* It will take approximately 15 to 30 minutes to answer the questions.

DETAILED DESCRIPTION:
In 2010, the Joint Commission (JC) issued a Sentinel Event Alert highlighting the need to detect suicide risk in all non-behavioral patients in medical settings. Detecting suicide risk among medical patients is important because this population is at elevated risk for suicidal thoughts and behaviors, and because for many of these patients, a medical visit is their only portal into mental health services. Of note, the vast majority of people who die by suicide visit a medical setting, such as an inpatient oncology unit, more frequently than a psychiatric setting in the months leading up to their death. Thus, the inpatient medical setting is an important stakeholder in decreasing suicide-related morbidity and mortality. Physicians and nurses working in non-mental health settings require tools to guide them in recognizing patients at risk. Nonetheless, there are currently no suicide screening instruments designed specifically for assessing suicide risk in an adult inpatient medical population.

In 2012, our study team conducted a Quality Improvement Project (QIP) at the National Institutes of Health Clinical Center (NIH CC) which demonstrated that the asQ em (Ask Suicide-Screening Questions to Everyone in Medical Settings), a brief instrument piloted to detect suicidal thoughts and behaviors among adult medical inpatients, was both feasible to administer and acceptable to both patients and staff. Extending this work, the aim of this current study is to further develop and psychometrically validate the asQ em among adult medical inpatients. While most inpatients will not be at imminent risk for suicide, we hypothesize that the asQ em will identify a number of patients who screen positive for suicide risk on a longer gold standard instrument, and that they are thus not only at risk for suicidal behavior in the future, but are also experiencing significant emotional distress and therefore warrant further mental health evaluation and recommendations for follow-up treatment.

This study will be a prospective, cross-sectional multisite study with patients enrolled from the NIH CC, Walter Reed National Military Medical Center, Rhode Island Hospital, and John Peter SmithHospital. The total planned sample size will be 810 (180 from WRNMMC, 180 from RIH, 200 from JPS, and 250 from NIH CC). We will administer several short measures of suicide risk: the 20 asQ em candidate items; a criterion standard Adult Suicidal Ideation Questionnaire (ASIQ); two questions which assess for suicidal behavior from a second criterion standard, the Beck Scale for Suicide Ideation (BSI); a brief depression screen, the Patient Health Questionnaire (PHQ-9); and an exploratory variable questionnaire, to all eligible inpatients aged 18 years and older. The ultimate goal of this project is the development of a validated risk of suicide screening instrument that can be administered rapidly by non-mental health clinicians to medical inpatients and in turn, connecting those in need with mental health services. Additionally, we hope to pilot the Suicide Implicit Association Test (S-IAT) in a subsample of recruited patients. The S-IAT is a brief computer task which measures a person s implicit association between self and either life or death . We expect to demonstrate that the S-IAT is feasible to administer in the inpatient medical setting thereby providing a potential alternative to self-report questionnaires for assessing patients thoughts about death or suicide.

Future studies will focus on examining the practical implications of nurses administering the asQ em as standard of care during the admission process on a medical inpatient unit and validating the asQ em in non-English speaking patients, addressing a critical gap in suicide prevention research. In addition, examining the long-term clinical impact of screening general medical patients for suicide risk with the asQ em and linking those in need with mental health services and/or other interventions will be important next steps.

ELIGIBILITY:
* INCLUSION CRITERIA:

All adult medical inpatients, ages 18 and older, who are admitted to selected medical units during data collection weeks will be approached for enrollment. Patients will be included if:

1. they are admitted as an inpatient on the designated medical units;
2. they are 18 and older;
3. they are capable of providing consent;

5) they have not previously been enrolled in this study.

EXCLUSION CRITERIA:

Patients will be excluded if:

1. they are medically or cognitively unable to participate in the screening or assessment (e.g., sustained altered level of consciousness, psychosis, hostile behavior, unremitting distress, intubation, persistent vomiting, severe pain, acute or worsening medical acuity);
2. they have been already enrolled during a previous visit;
3. they are unwilling to provide consent;
4. the patient is non-English speaking (because ASIQ has not been validated in languages other than English).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, cross-sectional multisite study. We will enroll adult patients, ages 18 years and older, admitted to identified inpatient medical units during designated data collections days. Patients will be recruited at the NIH CC as well as Walter Reed National Military Medical Center (WRNMMC), Rhode Island Hospital (RIH), and John Peter Smith Hospital (JPS).
Sampling Method: Non-Probability Sample
Enrollment: 740 (Actual)
Dates: Start 2014-05-14 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Short measures of suicide risk | Ongoing
  Short measures of suicide risk

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Horowitz, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (4):
- United States (4):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Rhode Island Hospital, Providence, Rhode Island
  - John Peter Smith Hospital, Fort Worth, Texas

REFERENCES:
- [Derived] Mournet AM, Bridge JA, Ross A, Powell D, Snyder DJ, Claassen CA, Wharff EA, Pao M, Horowitz LM. A Comparison of Suicide Attempt Histories of Pediatric and Adult Medical Inpatients and Implications for Screening. Arch Suicide Res. 2022 Jul-Sep;26(3):1541-1555. doi: 10.1080/13811118.2021.1931596. Epub 2021 Jun 8. PMID 34101537
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-M-0109.html